CLINICAL TRIAL: NCT04468087
Title: Antiviral for Adult Patients Hospitalized for SARS-CoV-2 Infection: a Randomized, Phase 2/3, Multicenter, Placebo Controlled, Adaptive, Multi-arm, Multi-stage Clinical Trial - Coalition Brazil COVID-19 IX: REVOLUTIOn
Brief Title: Antiviral Agents Against COVID-19 Infection
Acronym: REVOLUTIOn
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REVOLUTIOn
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: covid-19; antivirals; atazanavir; daclatasvir; sofosbuvir; multiarm multistage study; adaptive
MeSH Terms: conditions — COVID-19 | interventions — Atazanavir Sulfate; daclatasvir

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, multi-arm, multi-stage, study. Adults, COVID-19 confirmed by reverse-transcriptase-polymerase-chain-reaction (RT-PCR) or SARS-Cov2 Antigen hospitalized patients with ≤ 9 days duration of symptoms and SpO2<=94% will be randomly assigned to receive antivirals with potential effectiveness for SARS-CoV-2.
  The study is planned to be an adaptive phase II / III study. The phase II will be divided into 2 stages: first and second stages. First stage will allocate patients into a 3:3:3:1:1:1 allocation ratio (5 for each treatment group and 1 for placebo) and second stage will allocate into 2:2:1:1 (2 for each treatment group and 1 for placebo). The phase 3 study will then proceed in a 2:1 allocation (2 treatments for each placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study for participants of the same active drug and researchers. Both participant and investigator can know, after randomization, which medication they were allocated to. However, none will know whether the capsule to be administered is active or placebo, ensuring blinding within that specific group to which the participant was allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Atazanavir (Experimental): 600 mg (2 capsules) twice daily on the first day and 300 mg (1 capsule) twice daily for the subsequent 9 days.
  Interventions: Drug: Atazanavir
- Daclatasvir 60 mg (Experimental): initial dose of 120mg (2 capsules), followed by 60mg (1 capsule) once daily for 9 days.
  Interventions: Drug: Daclatasvir 60 mg
- Sofusbuvir + Daclatasvir 60 mg (Experimental): 400 mg twice daily (2 capsules) on the first day and 400 mg (1 capsules) once daily for the subsequent 9 days (sofosbuvir) + initial dose of 120mg (2 capsules), followed by 60mg (1 capsule) once a day for 9 days (daclastavir)
  Interventions: Drug: Sofusbuvir + Daclastavir 60 mg; Drug: Placebo Sofusbuvir + Daclatasvir 60 mg
- Placebo Atazanavir (Placebo Comparator): 2 capsules twice daily on the first day and 1 capsule twice daily for the subsequent 9 days.
  Interventions: Drug: Placebo Atazanavir
- Placebo Daclatasvir (Placebo Comparator): 2 capsules twice daily on the first day and 1 capsule twice daily for the subsequent 9 days.
  Interventions: Drug: Placebo Daclatasvir 60 mg
- Placebo Sofusbuvir + Daclatasvir (Placebo Comparator): 2 capsules twice daily on the first day and 1 capsule twice daily for the subsequent 9 days.
  Interventions: Drug: Placebo Sofusbuvir + Daclatasvir 60 mg

INTERVENTIONS:
Drug: Atazanavir — 600 mg (2 capsules) twice daily on the first day and 300 mg (1 capsule) twice daily for the subsequent 9 days.
  Other Names: Active Group
  Arms: Atazanavir
Drug: Daclatasvir 60 mg — initial dose of 120mg (2 capsules), followed by 60mg (1 capsule) once daily for 9 days.
  Other Names: Active Group
  Arms: Daclatasvir 60 mg
Drug: Sofusbuvir + Daclastavir 60 mg — 400 mg twice daily (2 capsules) on the first day and 400 mg (1 capsules) once daily for the subsequent 9 days (sofusbuvir) + initial dose of 120mg (2 capsules), followed by 60mg (1 capsule) once a day for 9 days (daclastavir)
  Other Names: Active Group
  Arms: Sofusbuvir + Daclatasvir 60 mg
Drug: Placebo Atazanavir — 2 capsules twice daily on the first day and 1 capsule twice daily for the subsequent 9 days.
  Other Names: Placebo group
  Arms: Placebo Atazanavir
Drug: Placebo Daclatasvir 60 mg — 2 capsules twice daily on the first day and 1 capsule twice daily for the subsequent 9 days.
  Other Names: Placebo group
  Arms: Placebo Daclatasvir
Drug: Placebo Sofusbuvir + Daclatasvir 60 mg — 2 capsules twice daily on the first day and 1 capsule twice daily for the subsequent 9 days.
  Other Names: Placebo group
  Arms: Placebo Sofusbuvir + Daclatasvir; Sofusbuvir + Daclatasvir 60 mg

SUMMARY:
A key strategy in the treatment of COVID-19 would be to find an effective antiviral agent that would decrease the peak viral load and, consequently, the associated degree of immunopathological damage that follows this phase. The clinically approved substances considered for this study are used for treatment of other virus diseases, like HIV (atazanavir) and HCV (sofosbuvir and daclatasvir). Severe progression of COVID-19 among patients under treatment for these aforementioned viruses is empirical less common. Besides, the clinical rationale, there are pre-clinical evidence pointing out that patients with COVID-19 could benefit from treatments with atazanavir, sofosbuvir and daclatasvir.

DETAILED DESCRIPTION:
We have planned an randomized, adaptive, placebo-controlled, double-blind study to be carried out in 3 seamless stages. The first two stages are phase 2 studies with a third stage phase 3 to be conducted conditional to success of the first phase 2 and second phase 2 stages including efficacy and safety.

In particular, there is great interest in the possibility of combining the phase II and phase III stages of the development process and this is the focus here. Phase II trials can be thought of as part of the learning stage where dose selection and appropriate treatment groups are assessed together with initial indications of their effects. Phase III trials are usually more confirmatory in nature where the treatment effects of the selected treatments are assessed in a full-scale trial. Seamless phase II/III trials are concerned with combining these two aspects into a single trial. There are a clearly advantages of speed in that the dose selection and treatment effects are assessed within a single trial rather than establishing separate trials. In addition, all data available for the selected dose are used in the analysis rather than just those from the second stage with a consequent gain in power. The savings in the number of patients is achieved by applying a form of screening of competing treatments in the initial phase and abandoning those that are ineffective before the end of the study following pre-established premises of futility. Effect estimates, confidence intervals and p values need some statistical adjustments to allow for this, otherwise they will be biased towards a benefit of the treatment. This study design, starting with a phase II, could give us a treatment regimen composed of one or more repurposed antivirals drugs that could improve the clinical outcomes of those hospitalized with COVID-19 reducing time to recovery and the need for respiratory support. It will be conducted in about 60 Brazilian hospitals.

Selection of drugs rationale

* Atazanavir: Atazanavir is a potent inhibitor of HIV-1 protease and is not associated with significant dyslipidemia, as observed with other protease inhibitors.15 It was approved by the FDA on January 29, 201516,17 as a combination of atazanavir and cobicistat. Atazanavir can also be combined with ritonavir18 In a protease-free cell assay, atazanavir blocked the major protease activity of SARS-Cov-2 at a concentration of 10 μM. In in vitro models of viral infection/replication performed on Vero cells, a human pulmonary epithelial cell line and primary human monocytes, atazanavir inhibited SARS-CoV-2 replication; in addition, the concentrations of interleukin 6 (IL-6) and tumor necrosis factor type alpha (TNF-α) induced by the virus were reduced.10 Currently, no clinical study is registered on the ClinicalTrials.com website to assess the effects of atazanavir in the context of COVID-19.
* Daclastavir: Daclatasvir is a direct-acting antiviral that inhibits HCV replication by binding to the N- terminal of the NS5A protein, affecting viral RNA replication. NS5A is a multifunctional protein in the HCV replicative cycle, involved in the enrollment of cell lipid bodies, RNA binding and replication, protein phosphorylation, cell signaling and antagonism of interferon pathways.19 In an in vitro study, daclatasvir consistently inhibited the production of SARS-CoV-2 infectious particles in Vero cells, in the HuH-7 cell line and in Calu-3 cells, with potencies of 0.8, 0.6 and 1.1 μM, respectively. Daclatasvir reached early events during the replication cycle of SARS-CoV-2 and prevented the induction of IL-6 and TNF-α, inflammatory mediators associated with the cytokine storm typical of SARS-CoV-2 infection.20
* Sofosbuvir/daclastavir:

Sofosbuvir (SOVALDI®) is a nucleotide analog directed against HCV NS5B polymerase, clinically approved with potent antiviral effects on the hepatitis C virus with several genotypes21. It is proposed that the drug could be a potential option in the treatment of COVID-19 especially at the beginning of the disease and before the invasion of the virus in the cells of the lung parenchyma, based on the similarity between the replication mechanisms of HCV and coronavirus22. In vitro, sofosbuvir showed EC50 values of 6.2 and 9.5 µM in HuH-7 (hepatoma) and Calu-3 (type II pneumocytes) cells respectively, although inactive in Vero cells (these cells are unable to make this conversion sofosbuvir in the pro-drug to active form)11.

First stage - will have 6 arms with total treatment for 10 days:

First stage Phase II - 6 arms

1. Atazanavir (ATV)
2. Daclatasvir (DCV)
3. Sofusbuvir+Daclatasvir (SFV/DCV)

6. Placebo (PbO) ATV 7. (PbO) DCV 8. (PbO) SFV/DCV

Second stage Phase II - 4 arms:

1. Best from first stage
2. Best from first stage + Second best
3. PbO Best from first stage;
4. PbO Best from first stage + Pbo Second best

Phase III - 2 arms:

1. Best from phase II second stage
2. (PbO) Best from phase 2 second stage

Main questions: The aim of the Coalition IX REVOLUTIOn evaluation is to answer the following questions:

* Are antiviral candidates (atazavir, daclatasvir/sofosbuvir) able to reduce the viral load of SARS-CoV-2 compared to placebo in patients hospitalized with COVID-19 with ≤ 9 days of symptoms?
* Which antiviral alone has the best effect in reducing the viral load of SARS-CoV-2 in patients hospitalized with COVID-19 with ≤ 9 days of symptoms? And which is the second most effective?
* Are combined antiviral candidates able to reduce the viral load of SARS-CoV-2 compared to antiviral alone and placebo in patients hospitalized with COVID-19 with ≤ 9 days of symptoms?
* Are isolated or combined antiviral candidates safe compared to placebo?
* Does the antiviral candidate alone or in combination improve clinical outcomes (days free of respiratory support in 15 days) compared with placebo in patients hospitalized with COVID-19 with ≤ 9 days of symptoms?

Primary/secondary objectives Primary objectives Phase II/ 1st and 2nd stages: Assess the effect of treatment with antivirals alone or combined with each other compared to placebo in reducing the of viral load of SARS-CoV-2 in nasopharyngeal swab samples obtained at baseline (d0) and days 3, 6 and 10; Phase III: Evaluate the effectiveness of best antivirals from Phase II alone or combined compared to placebo in increasing days free of respiratory support defined as the number of days without oxygen, non-invasive ventilation / high-flow nasal cannula or mechanical ventilation in 15 days.

Secondary Objectives

1. Ordinal 7-stage scale for clinical outcomes on the 15th day (1. not hospitalized with resumption of normal activities; 2. not hospitalized, but unable to resume normal activities; 3. hospitalized, without the need for supplemental oxygen; 4. hospitalized , requiring supplemental oxygen; 5. hospitalized, requiring high-flow nasal oxygen therapy, non-invasive mechanical ventilation or both; 6. hospitalized, requiring blood oxygenation through the membrane system, invasive mechanical ventilation or both; 7. Death);
2. Ordinal 6-stage scale for clinical outcomes on day 7 1. not hospitalized; 2. hospitalized, without the need for supplemental oxygen; 3. hospitalized, requiring supplemental oxygen; 4. hospitalized, requiring high-flow nasal oxygen therapy, non-invasive mechanical ventilation, or both; 5. hospitalized, requiring blood oxygenation through a membrane system, invasive mechanical ventilation or both; 6. Death;
3. Mortality in 28 days
4. Days free from mechanical ventilation within 28 days;
5. Days out of hospital within 28 days;
6. Time to discharge, defined as the number of days from randomization to discharge, within 28 days
7. Evaluate free days of respiratory support in 15 days for Phase II/1 and II/2
8. Grade 2, 3 or 4 adverse events that was not present at patient's admission, defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (corrected version 2.1, July, 2017); 53
9. Evaluate Serious adverse events (SAE);
10. Evaluate discontinuation of study drug-related treatment.

Recruitment and enrollment: The randomization list will be generated electronically using appropriate software. Randomization will be performed in blocks and stratified by center. The allocation concealment will be maintained through a centralized, automated, internet-based randomization system, available 24 hours a day. Hospitalized patients with the inclusion criteria will be allocated in an allocation ratio 3: 3: 3: 1: 1: 1 (3 for each treatment group and 1 for placebo) in Phase II / 1. The parameter of interest for the efficacy decision will be the comparison of the decay rates (slope) of the viral load logarithm from RT-PCR to COVID-19 in 10 days between the treatment groups in comparison with the control (placebo). In the 2nd stage, we will allocate patients in the ratio 2: 2: 1: 1 (2 for each active arm and 1 for each placebo) and the same statistic, now comparing combined treatment against the treatment selected in phase II / 1 and placebo, since it is already known that the treatment of phase II / 1 is effective for reducing viral load according to the pre specified criteria. As long as we have success on primary outcome of Phase II/2, Phase III will proceed in a 2: 1 allocation ratio (2 active treatments for each placebo).

Blinding:This is a double-blind study for participants of the same active drug and researchers. Both participant and investigator can know, after randomization, which medication they were allocated to. However, none will know whether the capsule to be administered is active or placebo, ensuring blinding within that specific group to which the participant was allocated.

Sample size and analysis: 252 patients in total in phase II first stage (189 in active groups and 63 in placebo) and 189 patients in total in phase II second stage (126 in active groups and 63 in placebo). In case of success in Phase II, 564 additional participants will be recruited in phase 3 (376 in the active group and 188 in the placebo). Thus, at the end of phase III, we will have 314 patients evaluated in the Placebo group and between 439 and 502 patients in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years) hospitalized with COVID-19:

   * SARS-CoV-2 positive RT-PCR or Antigen test
   * Typical clinical history and chest CT with typical findings, pending RT-PCR for SARS-CoV-2
2. Symptom duration <= 9 days
3. SpO2 <= 94% in room air or need for supplemental oxygen to maintain SpO2> 94%
4. The patient consents to participate in the study and is willing to comply with all study procedures, including the collection of virology samples

Exclusion Criteria:

1. Patients in need of respiratory support with invasive mechanical ventilation;
2. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal;
3. Total bilirubin > 2 mg/dL;
4. Platelets <50,000 cel/L;
5. Total neutrophil count <750 cell/L;
6. Renal dysfunction (estimated glomerular filtration rate [eGFR] <30 mL / min / 1.73 m2, using the MDRD or CKD-EPI method); and pre-defined renal failure stage 3 according to AKINx classification with serum creatinine> 4 mg / dl or patient already on renal replacement therapy;
7. Previously known liver disease (liver cirrhosis), defined as a report by the participant or written in the respective cirrhosis chart, esophageal varices, or the presence of clinical ascites on examination;
8. Decompensated congestive heart failure defined as the presence of dyspnea, edema of the lower limbs or rales on pulmonary auscultation, jugular turgency or chest X-ray with signs of pulmonary congestion;
9. Pregnant or breast feeding patients;
10. Known allergy or hypersensitivity to any study drug;
11. Hepatitis C carrier (HCV RNA positive), active Hepatitis B (positive surface antigen in the past), or HIV (ELISA and confirmatory Western Blot in the past). New screening tests are NOT required;
12. Patients currently using nucleoside or nucleotide analog drugs for any indication;
13. Corrected Q interval T> 480 on the electrocardiogram;
14. Heart rate <55 bpm;
15. Patients in use or who recently used (<90 days) amiodarone;
16. Women of childbearing potential and men with a partner of childbearing potential who do NOT agree to use two contraceptive methods (including barrier method) for 100 days.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Phase II first step: Change in the slope of SARS-COV 2 viral load | days 3, 6 and 10 after randomization
  Change in the slope of the SARS-COV 2 log viral load evaluated by nasopharyngeal swab samples assessed at baseline and days 3, 6 and 10 after randomization (isolated antiviral).
Phase II second step: Change in the slope of SARS-COV 2 viral load | days 3, 6 and 10 after randomization
  Change in the slope of the SARS-COV 2 log viral load curve evaluated by nasopharyngeal swab samples assessed at baseline and days 3, 6 and 10 after randomization (combined antiviral).
Phase III: Number of free days from respiratory support | 15 days
  Number of days without oxygen, non-invasive ventilation/high flow nasal cannula or need for mechanical ventilation in 15 days.

CONTACTS AND LOCATIONS:
Overall Officials: Israel S Maia, MSc, Principal Investigator — HCor Research Institute
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Maia IS, Marcadenti A, Veiga VC, Miranda TA, Gomes SPC, Carollo MBS, Negrelli KL, Gomes JO, Tramujas L, Abreu-Silva EO, Westphal GA, Fernandes RP, Horta JGA, Oliveira DC, Flato UAP, Paoliello RCR, Fernandes C, Zandonai CL, Coelho JC, Barros WC, Lemos JC, Bolan RS, Dutra MM, Gebara OCE, Lopes ATA, Alencar Filho MS, Arraes JA, Hamamoto VA, Hernandes ME, Golin NA, Santos TM, Santos RHN, Damiani LP, Zampieri FG, Gesto J, Machado FR, Rosa RG, Azevedo LCP, Avezum A, Lopes RD, Souza TML, Berwanger O, Cavalcanti AB; BRICNet. Antivirals for adult patients hospitalised with SARS-CoV-2 infection: a randomised, phase II/III, multicentre, placebo-controlled, adaptive study, with multiple arms and stages. COALITION COVID-19 BRAZIL IX - REVOLUTIOn trial. Lancet Reg Health Am. 2023 Apr;20:100466. doi: 10.1016/j.lana.2023.100466. Epub 2023 Mar 8. PMID 36908503
- [Derived] Maia IS, Marcadenti A, Zampieri FG, Damiani LP, Santos RHN, Negrelli KL, Gomes SPDC, Gomes JO, Carollo MBDS, Miranda TA, Santucci E, Valeis N, Laranjeira LN, Westphal GA, Horta JGA, Flato UAP, Fernandes C, Barros WC, Bolan RS, Gebara OCE, Alencar Filho MS, Hamamoto VA, Hernandes ME, Golin NA, Olinda RT, Machado FR, Rosa RG, Veiga VC, Azevedo LCP, Avezum A, Lopes RD, Souza TML, Berwanger O, Cavalcanti AB. Antivirals for adult patients hospitalized with SARS-CoV-2 infection: A randomized, Phase II/III, multicenter, placebo-controlled, adaptive study, with multiple arms and stages. COALITION COVID-19 BRAZIL IX - REVOLUTIOn: protocol and statistical analysis plan. Rev Bras Ter Intensiva. 2022 Jan-Mar;34(1):44-55. doi: 10.5935/0103-507X.20220002-pt. PMID 35766657